CLINICAL TRIAL: NCT03465098
Title: Evaluation of a Low-Carbohydrate Diet to Highlight Easily Infective Endocarditis by 18F-FDG PET
Brief Title: Evaluation of a Metabolic Preparation by a Low-carbohydrate Diet as Atkins-diet to Help in Detecting Infective Endocarditis by 18F-FDG PET
Acronym: TEPEIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Elodie CHEVALIER, Principal investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N°IDRCB: 2017-A01104-49
Record Dates: First submitted 2017-11-17; First posted 2018-03-14 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Infective Endocarditis
Keywords: Infective endocarditis; PET/CT 18F-FDG; Low carbohydrate diet as Atkins diet
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- enrolled patients (Experimental): All enrolled patients will be received a strict low carbohydrate (< 3gr/day of carbohydrate) and 12h fasting before 18F-FDG PET/CT exam and 24h after a 18F-FDG PET/CT preceded by a low carbohydrate diet with 12h fasting
  Interventions: Other: Strict low carbohydrate diet (< 3gr/day of carbohydrate) before a 18F-FDG PET/CT

INTERVENTIONS:
Other: Strict low carbohydrate diet (< 3gr/day of carbohydrate) before a 18F-FDG PET/CT — The patients will receive 2 PET/CT , first exam with standard diet preceded by 12h fasting and second exam preceded by 3 meals strict low diet and 12h fasting
  Other Names: 18F-FDG PET/CT

SUMMARY:
Infectious endocarditis (IE) is a pathology where the mortality rate of between 20 and 25%, but a higher morbidity since 50% of the patients are treated by a valvular surgical procedure. The diagnosis of IE is often difficult and therefore too late. In 2015, the European Society of Cardiology recommendations published by the integrate Positron Emission Tomography with Computed Tomography (PET/CT) with 18F-Fluorodeoxyglucose (18F-FDG) in the diagnostic management of IE.

However, during conventional examinations, with 12 hours fasting and low carb dieting, myocardial uptake of 18F-FDG may be intense and interfere with results.

The purpose of this study is to assess a strict low carbohydrate diet as Atkins (<3gram/day of carbohydrate) diet to facilitate the infective endocarditis diagnosis by 18F-FDG PET/CT Primary objective is to assess a strict low carbohydrate diet during 12h and 12h fasting for enhancing the contrast between infect area and surrounding structures and improve the detectability of infective endocarditis by PET/CT

Secondary objectives:

1. Comparison of the detection sensitivity of IE outbreaks between 18F-FDG PET/CT performed with the low carbohydrate diet and conventional diet performed
2. To assess the strict low carbohydrate diet effects on the uptake 18F-FDG distribution , particularly in the myocardium, circulating blood, skeletal muscles, brain and liver.
3. Characterization of metabolic changes generated by the low carbohydrate diet using plasma bioassays (blood glucose, insulinemia, free fatty acid concentration, ß-hydroxybutyrate).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with certainly infective endocarditis (95%) such Duke and Li criteria
* Patients with a social protection system
* No impossibility of performing (18)F-FDG PET (agitated, confused patient, etc)
* Stable clinically
* Adaptive antibiotic therapy for at least 8 days
* No known allergy to making impossible to follow strict carbohydrate diet

Exclusion Criteria:

* Pregnancy, breastfeeding and woman of childbearing age without effective contraception
* Patients under guardianship or curators.
* No treatment with corticoids, valproate, carbamazepine, phenytoin, phenobarbital, catecholamines
* Unbalanced diabetes (fasting capillary blood glucose > 1,8 g/l ou 10 mmol/l)
* Patients with known hypersensitivity to 18F-FDG or any component of this product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Infectious focus 18F-FDG activity measured with SUV (standardized uptake value ) | 24 hours
  The contrast will be measured thanks to the ratio SUV (standardized uptake value ) infectious focus and SUV (standardized uptake value ) surrounding tissue

SECONDARY OUTCOMES:
Visual analysis to detect and locate infective area | 24 hours
  each infectious focus will be appreciated by visual reading
SUV (standardized uptake value) of target organs (myocardium, muscles, liver, brain, blood, kidney..) | 3 days
  Measure of 18F-FDG activity on the target organs
metabolic biomarker assay: ß-hydroxybutyrate | one week (on PET standard and on PET with Atkins diet)
  impact diet on ß-hydroxybutyrate assay result (Measure of β-HydroxybutyrateB from plasma in µmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Elodie CHEVALIER, MD, Principal Investigator — Nuclear medicine department, CHRU NANCY
Locations (1):
- Chru Nancy Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No